CLINICAL TRIAL: NCT05517668
Title: A Randomized Controlled Study to Evaluate the Efficacy of Fomepizole in the Treatment of Acetaminophen Overdose
Brief Title: Evaluation of the Efficacy of Fomepizole in the Treatment of Acetaminophen Overdose
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Richard Dart, MD, PhD (Other)
Collaborators: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor-Investigator, Richard Dart, MD, PhD, Director RMPDS, Denver Health and Hospital Authority
Organization: Denver Health and Hospital Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-4745; 160034 (Other: FDA)
Record Dates: First submitted 2022-08-10; First posted 2022-08-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acetaminophen; Drug Overdose; Acetaminophen Overdose; Acetaminophen Poisoning; Drug-induced Liver Injury; Liver Failure; Liver Toxicity
MeSH Terms: conditions — Drug Overdose; Chemical and Drug Induced Liver Injury; Liver Failure | interventions — 4-methylpiperazine-2,6-dione

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (NAC) only (Control) (Active Comparator): Patients randomized to Control group will receive placebo (D5W) in addition to N-acetylcysteine. Study participants will receive study drug (fomepizole or placebo) throughout the study.
  Interventions: Drug: Intravenous infusion of N-acetylcysteine
- N-acetylcysteine (NAC) and Fomepizole (4-MP) (Study) (Experimental): Patients randomized to Study group will receive fomepizole (diluted in D5W) in addition to N-acetylcysteine. Study participants will receive study drug (fomepizole or placebo) throughout the study. If randomized to Study group, the infusion of the study medication should be initiated as soon as feasible but no later than 24 hours after the commencement of acetylcysteine therapy.
  Interventions: Drug: Intravenous infusion of N-acetylcysteine; Drug: Intravenous infusion of Fomepizole (4-MP)

INTERVENTIONS:
Drug: Intravenous infusion of N-acetylcysteine — If randomized to Control, the participant will receive only N-acetylcysteine. The dose will be determined by the site investigator. Typical continued infusion rate is 6.25 mg/kg/hr. The control drug (D5W) will be administered using the same schedule as fomepizole.
Drug: Intravenous infusion of Fomepizole (4-MP) — If randomized to fomepizole, the proposed infusion schedule for fomepizole closely mirrors the dosing outlined in the medication's package insert. Specifically, the Antizol (fomepizole) doses (bags) #1-5 allocated for the study will precisely adhere to the manufacturer's recommendations from the package insert. This entails an initial loading dose of 15 mg/kg followed by four subsequent doses of 10 mg/kg. The dose of fomepizole will not be adjusted based on age, presence of liver injury or renal insufficiency.
  Arms: N-acetylcysteine (NAC) and Fomepizole (4-MP) (Study)

SUMMARY:
This study is a randomized, placebo-controlled double-blinded clinical trial of patients presenting with acetaminophen poisoning who are at increased risk of developing liver injury. With this trial the investigators are hoping to show the superiority of acetylcysteine (NAC) + fomepizole (4-MP) compared to treatment with acetylcysteine alone. The primary objective of this trial is to determine the effect of fomepizole on the severity of acute liver injury in patients with acetaminophen poisoning.

DETAILED DESCRIPTION:
Acetaminophen (N-acetyl-p-aminophenol, paracetamol, APAP) is a commonly used analgesic and antipyretic. The maximal recommended therapeutic dose of 4 g per day is safe and is well tolerated. Unintentional and intentional overdoses occur and can cause serious hepatotoxicity. Acetaminophen overdose is the most common cause of drug-induced acute liver failure (ALF) in the US, accounting for 46% of all cases, which results in about 300-500 deaths annually. This is a persistent health problem because acetaminophen is widely available in the US market. Acetaminophen overdose can induce acute liver failure by a process that involves two processes: oxidative metabolism and amplification of oxidant stress.

Oxidative metabolism: At therapeutic doses, 95% of APAP is metabolized via glucuronidation and sulfation in the liver and eliminated from the body without resulting toxicity. In addition to these pathways, approximately 5% of an acetaminophen dose is metabolized by cytochrome P450 enzymes (mainly CYP2E1), which results in the formation of a highly reactive metabolite, N-acetyl-p-benzoquinone imine (NAPQI). During appropriate use of acetaminophen at therapeutic doses, the small amount of NAPQI produced is readily detoxified by intracellular glutathione. After an acetaminophen overdose, a much larger amount of acetaminophen is oxidized by CYP2E1 resulting in elevated amounts of NAPQI. When the amount of NAPQI generated exceeds hepatic glutathione stores, NAPQI binds to cellular and mitochondrial proteins causing dysfunction. This cascade can be amplified through other mediators leading to DNA damage and hepatocyte death.

Amplification of oxidant stress: After NAPQI formation, c-Jun N-terminal kinase (JNK) activation in the cytosol of the cell and its mitochondrial translocation results in the induction of the mitochondrial membrane transition pore. This ultimately triggers a molecular cascade causing amplification of mitochondrial oxidant stress, nuclear DNA fragmentation, and hepatic cell death.

Acetylcysteine is the only FDA approved drug indicated for clinical use in acetaminophen overdose. It is highly effective when patients seek medical attention within 8 hours of acute single ingestion. The incidence and severity of clinically important liver injury after acute ingestion of acetaminophen increases when acetylcysteine is started over 8 hours after ingestion. Many patients, however, seek medical attention later, when acetylcysteine has reduced efficacy thus putting some patients at risk of developing hepatotoxicity, fulminant hepatic failure and death despite acetylcysteine therapy. While not a frequent occurrence, the effects are devastating to the patient and their family. Acetylcysteine acts by replenishing reduced glutathione, but it only addresses the oxidative phase of acetaminophen toxicity. A novel therapeutic intervention strategy is needed for the treatment of acetaminophen-induced hepatotoxicity in these higher risk patients.

Fomepizole (4-methylpyrazole) is an FDA approved medication for the treatment of patients with toxic alcohol poisoning by blocking the activity of alcohol dehydrogenase. However, fomepizole has other effects. In animal models of acetaminophen poisoning, fomepizole has been demonstrated to inhibit both phases of acetaminophen-induced liver injury: oxidative metabolism and amplification of injury through JNK and other mediators. Also, inhibition of JNK activation and its resulting mitochondrial translocation and amplification of mitochondrial oxidant stress has been shown to prevent acute liver injury in animal studies. Therefore, fomepizole appears to work in two ways: protection early in the course by preventing the oxidative metabolism of acetaminophen to NAPQI through inhibition of CYP2E1. Additionally, it is important to note that it appears protective late in the clinical course after NAPQI has been formed by inhibiting JNK activation and preventing cell death.

The investigators propose fomepizole as an adjunctive therapy to acetylcysteine because it adds two additional mechanisms of action, has been studied in the appropriate animal models, and off-label use in humans is promising. Acetylcysteine improves the redox environment is the cell by fostering the regeneration of reduced glutathione (GSH). Fomepizole complements this mechanism by reducing metabolism of acetaminophen to NAPQI, thereby greatly reducing the initial stimulus to injury. In addition, it reduces activation of JNK, which reduces amplification of the injury initiated by NAPQI. Fomepizole therapy is expected to have significant value in patients who are at increased risk of liver injury despite treatment with acetylcysteine. Today, nearly all deaths from acetaminophen arise from this group.

A randomized controlled trial (RCT) was chosen as the strongest type of trial to assess efficacy of Fomepizole. The investigators could potentially have used a single arm study and used historical controls. However, the evolution of acetaminophen treatment in recent years as well as the increasing incidence of patients with repeated supratherapeutic ingestions (RSTI) indicates that it is preferable to have a contemporaneous comparison group.

An inactive control was chosen because current treatment of acetaminophen poisoning is well characterized and there are no other plausible antidotes other than acetylcysteine available to provide an active comparator.

The investigators have included both acute and repeating ("chronic") patterns of acetaminophen ingestion for several reasons. The main reason is that the clinical reality of acetaminophen poisoning is that many patients don't accurately report the pattern or amount of their ingestion. A prospective assessment of clinician confidence in the acetaminophen dose or time of last ingestion found that physicians were confident in the history in only 16.7% of cases involving acute ingestion of acetaminophen and 0% of cases involving chronic overdose. An ingestion of acetaminophen is often combined with other agents such as alcohol and thus their recollection of events is often inaccurate. Often a patient who claims they took a single acute ingestion is inaccurate. They may view their ingestion as acute, but actually ingested the tablets over many hours. Others take an acute ingestion on the background of overuse of the acetaminophen. Still others repeatedly take supratherapeutic doses for multiple days. It would be impossible to parse these patients for enrollment because even a detailed history would provide myriad and often inaccurate information.

Fortunately, the published medical literature and our own experience in off-label use of acetylcysteine suggest that fomepizole's mechanism of action should be effective in all patterns of ingestion. However, there is one scenario where fomepizole (or any treatment) will be ineffective - patients whose injury has progressed so far that only liver transplant offers hope. Therefore, the investigators plan to exclude the group of patients that present with advanced injury that is unlikely to respond to treatment.

Each patient will receive acetylcysteine treatment throughout their hospitalization. Clinical toxicologists in US use a relatively common definition of when to stop treatment every 12 hours after initiation of acetylcysteine. Infusion of acetylcysteine is terminated when all the following conditions ("Stopping Rule" are met):

1. the patient's serum acetaminophen has become undetectable (less than 10 mg/L),
2. ALT/AST levels are considered normal for the patient, or if elevated, at least one of them (either ALT or AST) has decreased from its peak by at least 25%,
3. the INR (international normalized ratio) is below 2.0, and
4. the patient is clinically well.

Both acetylcysteine and study drug will be terminated when this criterion is met. Study drug will be terminated after 5 days (120 hours) after initiation of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of acute or repeated supratherapeutic ingestion (RSTI)* of acetaminophen (serum acetaminophen greater or equal to 10 mg/L) after correction for bilirubin, when applicable**
2. Baseline AT Multiplication Product at screening ([APAP] multiplied by the serum AST or ALT in IU/L, whichever is higher) of 3000 or higher
3. Adults and children ages 10 years or older
4. Infusion of NAC started 8 hours or more post-ingestion
5. Infusion of the study medication begins as early as possible but not later than 24 hours after the initiation of the NAC infusion.
6. Patient presenting to or transferred to the participating site hospital and planned to be admitted to hospital for treatment and/or observation or treatment in Emergency Department
7. Provision of signed and dated informed consent form
8. Stated willingness to comply with mandatory study procedures and availability for the duration of the study

Exclusion Criteria:

1. Serum ALT greater than 10,000 IU/L or serum AST greater than 20,000 IU/L at time of screening
2. Another overdose episode with acetaminophen within the preceding 14 days
3. Baseline ALT (defined as average of ALTs reported in preceding 12 months) above the ALT reference range for the hospital laboratory unless screening ALT is at least twice the patient's baseline value.
4. Evidence of chronic decompensated liver cirrhosis regardless of serum ALT activity***
5. Known allergic reaction to acetylcysteine or a documented serious hypersensitivity reaction to fomepizole or other pyrazoles.
6. Pregnancy or lactation
7. Co-ingestion of other known activators or inhibitors of CYP2E1 (acetone, cimetidine, nicotine, isoniazid, pyridine, pyrazole, disulfiram). History of cigarette smoking, use of nicotine patches are allowed.
8. Concomitant ingestion of high dosage iron preparations (e.g., prenatal iron sulfate capsules)
9. In the site investigator's judgment, the patient has a condition that would interfere with evaluation of the efficacy of fomepizole. These conditions include, but are not limited to the following conditions:

   * Seizure in the previous 24 hours. History of seizure disorder under chronic treatment is allowed
   * Cardiac arrest in the preceding 14 days
   * Cardiac dysrhythmia that compromises cardiovascular function at screening
   * History of liver transplant
   * Shock liver
10. Treatment with another investigational drug within the preceding 30 days.
11. Previous participation in this study

    * Acute ingestion is defined as more than 4 grams ingested over 24-hour period. RSTI defined as more than 4 grams ingested/24 hour period for more than 24 hours. Note: the type of ingestion (acute vs. RSTI) or its timing relative to time of hospital admission do not affect neither study eligibility nor research subject management.

      * Bilirubinemia (high bilirubin in blood) may cause falsely elevated APAP levels when tested with spectrophotometric assay (SPA). In order to rule out this false elevation we recommend validating APAP level via liquid chromatography (LC) or mass spectrometry (MS) testing methods after we enroll a patient with APAP test results between 10 and 30 mg/L and total bilirubin ≥ 10 mg/dL.

        * Decompensated cirrhosis refers to a stage of liver cirrhosis where the liver is no longer able to function properly due to extensive damage, scarring, and fibrosis. Patients with decompensated cirrhosis may have symptoms such as jaundice (yellowing of the skin and eyes), ascites (abdominal swelling), gastrointestinal bleeding, spider angiomas (red, spider-like lesions on the skin), hepatic encephalopathy (confusion and cognitive impairment), or hepatorenal syndrome (kidney dysfunction). Decompensated cirrhosis is a more advanced and serious stage of liver disease, and patients may require hospitalization and more aggressive medical interventions, including liver transplantation.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
Difference in serum alanine transaminase (ALT) from presentation to peak recorded ALT | ALT will be measured at baseline, then at 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Determine the effect of fomepizole on the severity of acute liver injury in patients with acetaminophen ingestion. Serum ALT is a recognized measure of liver injury. A smaller increase in ALT indicates the efficacy of the study drug.

SECONDARY OUTCOMES:
Time to meet endpoints for termination of acetylcysteine infusion | Study participants will be evaluated for study medication discontinuation at 12, 20, 32, 44, etc. hours after starting NAC (every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Determine effect on clinical practice. Shorter time to endpoint indicates improved efficacy compared to treatment with acetylcysteine alone.
Peak INR | INR will be measured at baseline, then at 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Determine the effect of fomepizole on other measures of liver injury and acute liver failure. INR is a measure of hepatic function.
Peak aspartate aminotransferase (AST) | AST will be measured at baseline then at 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Determine the effect of fomepizole on other measures of liver injury and acute liver failure. AST is a measure of hepatic injury.
Peak creatinine | Creatinine will be measured at baseline then at 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Determine the effect of fomepizole on measures of kidney injury. Creatinine is a measure of kidney injury.
Measurement of protein adducts | Protein adducts will be measured at 2, 5, 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Assess contribution of CYP2E1 inhibition by fomepizole effect, if any. Decreased protein adduct concentration in blood indicates fomepizole has blocked CYP2E1.
Proportion of patients developing acute liver failure (ALF). | INR, ALT and AST will be measured at baseline, then at 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Assess overall incidence of acute liver failure (ALF).
Serial measurement of fomepizole serum concentration | Fomepizole serum concentration will be measured at 2, 5, 12, 20, 32, 44, etc. hours after starting NAC (and every 12 hours afterwards) as long as patient is receiving medication (either NAC or NAC and 4-MP), two to three days on average.
  Assess pharmacokinetic profile of fomepizole. Assess whether continuous infusion produces steady concentration.

OTHER OUTCOMES:
Measurement to perform a candidate gene analysis of CYP2E1, glutathione synthetase, UDP-glucuronosyltransferases, JNK related to APAP toxicity. | Pharmacogenomics will be measured at 5 hours after study subject starts receiving NAC.
  Determine genetic variants of acetaminophen overdose and response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dart, MD, PhD, Principal Investigator — Rocky Mountain Poison and Drug Safety, division of Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No